CLINICAL TRIAL: NCT01916811
Title: Load Quantitative MRI Study of Incipient LBP Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Hongbin Lu, Professor, Central South University
Other Study IDs: 20130114
Record Dates: First submitted 2013-08-03; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Load quantitative MRI
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The mian purpose of this study is to analysis the imaging changes in 3.0T MRI of lumbar small joints, intervertebral discs, ligaments and muscle in hospital nurses first suffered with low back pain.

DETAILED DESCRIPTION:
Low back pain is a common clinical disease seriously affects the quality of people's lives. And this disease takes up a large proportion in the crowd. Incipient lumbago is hard to diagnose and often hidden morbidity. If early symptoms are ignored by patients, it will greatly influence the quality of life in the future. This study will use 3.0T MRI to distinguish the difference of lumbar small joints, intervertebral discs, ligaments and muscle between the normal and the pain.

Firstly, we recruit nurses with low back pain in one group, with the normal as control. Then the subject will accept 3.0T MRI scanning at the same time. Before scanning we will determine the MRI sequence to make sure the imageis are clear enough. At last, we will analysis the photos in the image processing workstation, reconstruct the anatomical structure in the scanning area. All of this is to find a possible reason or explanation in the occurrence of incipient lumbago through the comparison of two group's images.

ELIGIBILITY:
Inclusion Criteria:

1. Female between 18 and 27 years of age
2. Subject who has worked as a nurse less than three years and will continue working as a nurse no less than one year
3. Back pain has happened more than 2 times In the past 12 months(every time lasts 2 days or more),or never happened
4. Subjects who do not participate any other study concerning pain prevention currently and in the next year
5. According with magnetic resonance inspection standard
6. NO spectical low back pain and no other serious diseases in the other systems

Exclusion Criteria:

1. Subjects who has a family history of low back pain
2. Subjects who are Suffering from specific low back pain
3. Subjects who are suffering from serious somatic disease and/or psychic disease
4. Subjects who are suffering from chronic pain disease and need long-term use of drug therapy
5. Subjects who are pregnant, planning to have a baby in 1 year or less than 6 months after delivery
6. Subjects who are suffering from chronic cardiac, respiratory, liver and kidney complaint symptomatically
7. Subjects who have had a spinal operation

Ages: 18 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young female nurse
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
the structure of lumbar | 18 months
  research the structure of facet joint,disc,muscle and ligment using quantitative MRI.

SECONDARY OUTCOMES:
the function of lumbar | 18 months
  research the function of facet joint,disc,muscle and ligment using quantitative MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hongbin, M.D. & Ph.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China